CLINICAL TRIAL: NCT06244589
Title: Evaluation of Risk Factors Leading to Conversion From Laparoscopic Cholecystectomy to Open Surgery: A Retrospective Controlled Study
Brief Title: Evaluation of Risk Factors Leading to Conversion From Laparoscopic Cholecystectomy to Open Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Burak Dincer, Burak Dinçer, MD, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16.01.2024-4240
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Cholelithiasis; Cholecystitis, Acute; Cholecystitis, Chronic; Gallbladder Diseases
Keywords: Laparoscopic cholecystectomy; Conversion; Cholelithiasis; Acute cholecystitis
MeSH Terms: conditions — Cholelithiasis; Cholecystitis, Acute; Cholecystitis; Bronchiolitis Obliterans Syndrome; Gallbladder Diseases | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: The study aims to compare cases of laparoscopic cholecystectomy with those undergoing open-conversion cholecystectomy to assess factors influencing the conversion to open surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic cholecystectomy (Active Comparator): Cases that laparoscopic cholecystectomy performed without need for open-conversion
  Interventions: Procedure: Laparoscopic cholecystectomy
- Open-conversion cholecystectomy (Experimental): Cases converted to open surgery based on intraoperative findings.
  Interventions: Procedure: Laparoscopic cholecystectomy; Procedure: Open-conversion cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy: Cholecystectomy that performed with laparoscopic method
Procedure: Open-conversion cholecystectomy — Open-conversion cholecystectomy: Cases in which laparotomy (Generally right subcostal incision) was performed based on intraoperative findings.
  Arms: Open-conversion cholecystectomy

SUMMARY:
This retrospective controlled study aims to evaluate risk factors that affect open conversion in laparoscopic cholecystectomy. Patient characteristics, medical history, biochemical and radiological studies of the patient will searched from the hospital database and factors affecting open conversion will be analysed.

DETAILED DESCRIPTION:
Cholecystectomy is a commonly performed procedure in general surgical practice, and with advancements in technology, it is widely conducted using the laparoscopic method. Despite the decreasing trend in open surgical procedures with increasing experience and technological developments, the literature reports conversion to open surgery in laparoscopic cholecystectomy ranging from 2% to 15%. Although some studies exist regarding patient groups at risk of conversion to open surgery, the current literature is insufficient to draw a clear conclusion on this matter. This study aims to evaluate risk factors for conversion to open surgery by examining cases of laparoscopically initiated cholecystectomy.

The study will be conducted retrospectively by reviewing archive records. Patients operated for cholecystectomy will be included. Patients that open surgical method used from start will be excluded from study. Age, comorbidities (ASA score), laboratory findings (leukocyte count and CRP), imaging findings (abdominal ultrasound, CT, or MRI), history of previous abdominal surgery, history of ERCP, and history of pancreatitis will be evaluated. Laparoscopic cholecystectomy cases will be compared with open-conversion cholecystectomies to assess factors influencing the conversion.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 95 years old.
* Operated for gallbladder disease (Cholecystectomy)
* Surgery must started with laparoscopic approach

Exclusion Criteria:

* Open surgery from the start
* Cholecystectomy as a part of bigger surgical intervention (Such as pancreaticoduodenectomy)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1695 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Open-conversion rate | Immediately after the surgery
  The rate of cases converted to open surgery among all laparoscopic cholecystectomy cases.

SECONDARY OUTCOMES:
Postoperative complication rate | 1 months after the surgery
  The rate of postoperative complications
Incidental gallbladder malignancy rate | 1 months after the surgery
  The rate of incidentally diagnosed gallbladder cancer among all laparoscopic cholecystectomies in patients without a preoperative diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Dincer, M.D., Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dincer B, Omeroglu S, Tufan AE, Uzun MA. Evaluation of Risk Factors Leading to Conversion from Laparoscopic Cholecystectomy to Open Surgery: A Retrospective Controlled Study. J Laparoendosc Adv Surg Tech A. 2025 Mar;35(3):204-209. doi: 10.1089/lap.2024.0366. Epub 2025 Feb 24. PMID 39992726